CLINICAL TRIAL: NCT04238091
Title: Open Label Clinical Trial to Evaluate the Efficacy of Fecal Microbiota Transplantation in Patients With Alopecia Areata
Brief Title: Clinical Trial to Evaluate the Efficacy of Fecal Microbiota Transplantation in Patients With Alopecia Areata
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator is no longer interested in moving forward with this study
Sponsor: Lindsey Bordone (Other)
Responsible Party: Sponsor-Investigator, Lindsey Bordone, Assistant Professor of Dermatology, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS4183
Record Dates: First submitted 2020-01-14; First posted 2020-01-23 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis
Keywords: Hair Loss; Alopecia
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis; Alopecia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Antibiotics prior to FMT (Active Comparator): Participants will take a standardized regimen of antibiotics for three days prior to fecal transplant.
  Interventions: Drug: Fecal material transfer therapy; Procedure: 4mm Punch Biopsy of Scalp; Diagnostic Test: Blood draw; Procedure: Skin Microbiome sampling; Procedure: Hair Microbiome Sampling; Drug: Pre-FMT Antibiotic Cocktail; Drug: Bowel Prep
- No Antibiotics prior to FMT (Active Comparator): Participants will not take antibiotics before the transplant.
  Interventions: Drug: Fecal material transfer therapy; Procedure: 4mm Punch Biopsy of Scalp; Diagnostic Test: Blood draw; Procedure: Skin Microbiome sampling; Procedure: Hair Microbiome Sampling; Drug: Bowel Prep

INTERVENTIONS:
Drug: Fecal material transfer therapy — Fecal microbiota transplants will be performed as follows:
  FMP Retention Enema: (FMP 250 mL) Dosage Form: Screened human donor stool, suspended in diluent of 12.5% glycerol and sterile normal saline buffer (0.9% NaCl) standardized to a 5X concentration (1g stool : 5mL diluent ratio), homogenized, filtered to 330 microns and aliquoted to sterile 250mL vessels.
  Route of Administration: Fecal transplant will be performed under medical supervision. Lubricated enema tube will be inserted into rectum and contents expelled into the distal colon with the subject requested to retain material for a target dwell time of 3 to 24 hours with a mean target of 10 hours. Participants will lie in the left lateral decubitus position but if mobility permits will rotate to supine and right lateral decubitus position.
  One half of study subjects will receive a 3 day course of antibiotics prior to fecal transplant, while the other half will not.
  Other Names: FMT
Procedure: 4mm Punch Biopsy of Scalp — For the skin biopsy, the doctor will select an appropriate area on the scalp (or skin) as the biopsy site. The area will then be numbed (anesthetized). The study doctor or his/hers designee will then use a cylindrical instrument with a sharp edge (similar to a small cookie-cutter) to remove a 4mm cylinder of skin (smaller than the size of a pencil eraser). After the skin is removed, the biopsy site will be closed with absorbable stitches when appropriate. Approximately 2 to 4 stitches may be placed at the wound site to improve healing. Multiple skin punch biopsies may be taken throughout the entire length of the study
  Other Names: Punch Biopsy of Scalp
Diagnostic Test: Blood draw — Blood will be collected by a standard venipuncture procedure. 60-80cc of blood will be drawn from a patient per blood draw occurrence. Blood samples will be transferred to the research facility. Samples will be used to either stained with cell surface antibodies for fluorescence acquisition cell sorting (FACS) analysis (FACS experiments will allow for assessment of the subset and activation status of immune cells involved in AA or other cutaneous disorder pathology) or to extract DNA for the purposes of exome or genomic sequencing or genotyping of disease associated genes
Procedure: Skin Microbiome sampling — Skin microbiome will be collected using skin swabs at the time of recruitment according to established protocols outlined by the Human Microbiome Project. Sterile (germ-free) techniques will be used for collection of all specimens, with careful avoidance of contamination of collection area by gloved hands. The sites that will be sampled are (in sequence): Lesional AA skin, non-lesional scalp skin, retro-auricular crease, ante-cubital fossa, and anterior nares. Skin surface specimens will be collected with a Catch-All Sample Collection Swab swab that looks similar to a q-tip and is, moistened with sterile solution. Skin will be swabbed approximately 50 times along the scalp, behind your ear and on your arm, and twisted 2 times around the front of the nose.
Procedure: Hair Microbiome Sampling — Hair follicle microbiome (bacteria that live in the hair follicle) will be collected as follows: several hairs will be plucked from the scalp at a time using tweezers, once plucked the bulbs of the hairs will be cut using sterile surgical scissors and processed. Approximately 10-15 hairs will be plucked for processing. The number of hairs plucked may be increased depending on the number of hairs containing bulbs. Up to 50 hairs may be plucked, as long as the subject is able to tolerate it. Only several hairs will be plucked at a time in order to minimize pain and discomfort of the procedure.
Drug: Pre-FMT Antibiotic Cocktail — For three days prior to the transplant, one half (20) of the subjects enrolled will be treated with antibiotics to reduce the burden of the existing microbiome. The antibiotic regimen will consist of: oral vancomycin 250 mg qid, ciprofloxacin 500 mg bid, and metronidazole 500 mg tid. For subjects who have antibiotic allergies, appropriate antibiotic substitutions will be made. Subjects will stop the antibiotics 48 hours before the fecal transplant.
  Arms: Antibiotics prior to FMT
Drug: Bowel Prep — The night before the transplant, all enrolled subjects will take 20 mg of bisacodyl and a large volume bowel preparation (GoLyteley 4000cc). Fecal transplant will be performed under medical supervision. After the transplant, subjects will take 4 mg of loperamide to increase transplant retention.

SUMMARY:
The purpose of this study is to examine fecal transfer as a potential treatment for Alopecia Areata (AA). This trial will attempt to discover if fecal transfer can treat immune-related hair loss.

DETAILED DESCRIPTION:
Alopecia areata (AA) is an autoimmune condition resulting in chronic and relapsing hair loss. AA patchy is associated with well-circumscribed patches of hair loss, commonly on the scalp or face, while alopecia totalis (AT) and alopecia universalis (AU) are two severe types of AA characterized by 95% or more hair loss on the scalp (AT) or body (AU). Although the exact underlying mechanisms that cause AA are unknown, T lymphocyte cells are implicated, as they release pro-inflammatory cytokines and chemokines around the hair follicles, triggering a cascade and ultimately resulting in hair loss.

Fecal microbiota transfer (FMT) involves the transfer of stool (feces) from a healthy donor to an AA recipient. Research suggests that changing the type of bacteria in an individual's intestine may carry the potential to alter (increase or decrease) the recipient's potential for certain conditions, even autoimmune conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 75 years of age with moderate to severe alopecia areata (SALT score >30%)
* Patients with a diagnosis of patch type alopecia areata, totalis, or universalis.
* Duration of hair loss greater than 3 months.
* No evidence of active, ongoing regrowth present at baseline.
* Females of childbearing potential must have a negative urine or serum pregnancy test at screening and immediately prior to FMT on the day of FMT, and
* Females of childbearing potential must agree to use an effective form of contraception from 14 days prior to study antibiotics through at least 30 days after FMT. Acceptable forms of contraception include Oral/intramuscular (IM) contraceptives, intrauterine device (IUD), surgical sterilization.

Exclusion Criteria:

* Inability (e.g. dysphagia) to or unwilling to swallow capsules
* Active gastrointestinal infection at time of enrollment
* Patient received antibiotics in the last 48 hours. Patients will be eligible to enroll if antibiotic therapy is discontinued for at minimum 48 hours prior to treatment.
* Requires continued antibiotic use or anticipates antibiotic use in the upcoming 4 weeks
* Known or suspected toxic megacolon and/or known small bowel ileus
* Major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment. This does not include appendectomy or cholecystectomy
* History of total colectomy or bariatric surgery
* Concurrent intensive induction chemotherapy, radiation therapy or biological treatment for active malignancy
* Unable or unwilling to comply with protocol requirements
* Expected life expectancy < 6 months
* Previous FMT or microbiome-based products at any time excluding this study
* Patients with a history of severe anaphylactic or anaphylactoid food allergy
* Solid organ transplant recipients 90 days post-transplant or on active treatment for rejection
* If at risk for CMV/EBV associated disease (at investigator's discretion, e.g. immunocompromised), negative immunoglobulin G (igG) testing for cytomegalovirus (CMV) or Epstein Barr Virus (EBV).
* A condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the results of the study
* Patients with a history of or existing skin diseases affecting the scalp such as psoriasis or seborrheic dermatitis and patients with evidence of infection or skin cancer in the treated areas
* Patients in whom the diagnosis of alopecia areata is questionable
* Patients in whom regrowth is present/evident at baseline in the areas to be treated
* Patients with active medical conditions or malignancies (except adequately treated basal or squamous cell carcinoma of the skin) which in the opinion of the investigator would increase the risks associated with study participation, including patients with a history of recurrent infections
* Patients known to be HIV or hepatitis B or C positive or otherwise immunocompromised
* Patients unwilling or unable to discontinue treatments known to affect hair regrowth in alopecia areata
* Patients who have been treated with intralesional steroids, systemic steroids, anthralin, squaric acid, diphenylcyclopropenone (DPCP), protopic, minoxidil, Janus kinase (JAK) inhibitors or other medication which in the opinion of the investigator may affect hair regrowth, within one month of the baseline visit.
* Patients determined by the investigator to have extreme diets.
* Patients (children) under the age of 18.
* Pregnant and breastfeeding females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Number of responders in patients treated with FMT | 24 weeks post-treatment
  Responders are defined as subjects achieving 50% or greater (% change, NOT absolute change) hair re-growth from baseline as assessed by SALT (Severity of Alopecia Tool) score where 0 indicates no hair and 100 is a full head of hair (i.e. 50% regrowth at week 24). A higher SALT score/ higher percent change indicate a better outcome.
Proportion of participants with an adverse event (AE) through day 30 (±3 days) after FMT | 30 days post-treatment
Proportion of participants with a serious adverse event (SAE) through day 30 (±3 days) after FMT | 30 days post-treatment
Proportion of participants with newly acquired transmissible infectious diseases which are considered adverse events of special interest (AESI) through day 30 (±3 days) after FMT | 30 days post-treatment

SECONDARY OUTCOMES:
Time of relapse in responders | 24 weeks post-treatment
  The timing of relapse in responders will be followed for 6 months post therapy.
Proportion of participants with an AE through week 4 (±5 days) after FMT | 4 weeks post-treatment
Proportion of participants with an SAE through week 4 (±5 days) after FMT | 4 weeks post-treatment
Proportion of participants with a SAE at month 6 (±14 days) after randomization | 6 months post-randomization
Proportion of participants with a SAE at month 12 (±14 days) after randomization | 12 months post-randomization
Percent hair regrowth from baseline | 24 weeks post-treatment
  This will be determined by SALT measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Bordone, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie WR, Yang XY, Xia HH, Wu LH, He XX. Hair regrowth following fecal microbiota transplantation in an elderly patient with alopecia areata: A case report and review of the literature. World J Clin Cases. 2019 Oct 6;7(19):3074-3081. doi: 10.12998/wjcc.v7.i19.3074. PMID 31624757
- [Background] Rebello D, Wang E, Yen E, Lio PA, Kelly CR. Hair Growth in Two Alopecia Patients after Fecal Microbiota Transplant. ACG Case Rep J. 2017 Sep 13;4:e107. doi: 10.14309/crj.2017.107. eCollection 2017. PMID 28932754